CLINICAL TRIAL: NCT04306913
Title: Outcome of Esmolol Potassium Cardioplegia Compared to Potassium Cardioplegia in Patients With Solitary Valvular Disease; Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, Consultant, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D-47-2019
Record Dates: First submitted 2020-03-02; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cardioplegia Solution Adverse Reaction
MeSH Terms: interventions — esmolol; potassium cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Potassium Cardioplegic Solution
- Esmolol (Experimental)
  Interventions: Drug: Esmolol; Drug: Potassium Cardioplegic Solution

INTERVENTIONS:
Drug: Esmolol — esmolol 250 mg in cardioplegia solution every 25 minutes
  Arms: Esmolol
Drug: Potassium Cardioplegic Solution — 15 meq potassium added to cardioplegia solution

SUMMARY:
Perioperative myocardial injury remains one of the most serious complications of cardiac surgery.

Numerous factors have been implicated during the pathogenesis process, including the technique of cardiac surgery, induction of cardioplegia and period of cardiac arrest.

Lactic acid is the normal endpoint of the anaerobic breakdown of glucose in the tissues. The lactate exits the cells and is transported to the liver, thus it's considered to be an indicator of ischemia as it is produced by most tissues in the human body, with the highest level of production found in muscle.

In any cardiac valve replacement surgery, patient must undergo cardiac bypass and arrest in diastole by using hyperkalemic cardioplegia solution; meanwhile the metabolism of myocardial cells is purely anaerobic.

Esmolol an ultra-short beta blocker is supposed to decrease the anaerobic insult to the myocardial cells.

ELIGIBILITY:
Inclusion Criteria:

- 20-50 years old patients, with either sex with solitary valvular disease

Exclusion Criteria:

* • Myocardial infarction within 2 weeks.

  * History of reaction or toxicity to esmolol or other beta blockers.
  * New York Heart Association class IV congestive heart failure despite treatment.
  * Persistent hypotension (systolic blood pressure <80 mm Hg).
  * severe pulmonary hypertension
  * Ejection fraction less than 45%
  * Patients with coronary artery disease
  * Patients with congenital heart disease
  * Patients with previous cardiac surgery
  * Patients with liver disease (child class B and C)
  * Patients with second or third degree heart block
  * Patients having resting heart rate less than 50 ppm
  * Patients using calcium channel blockers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Coronary sinus lactate level immediately before declamping the aorta. | 1 hour during declamping
  the lactate from the coronary sinus

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scorsin M, Mebazaa A, Al Attar N, Medini B, Callebert J, Raffoul R, Ramadan R, Maillet JM, Ruffenach A, Simoneau F, Nataf P, Payen D, Lessana A. Efficacy of esmolol as a myocardial protective agent during continuous retrograde blood cardioplegia. J Thorac Cardiovasc Surg. 2003 May;125(5):1022-9. doi: 10.1067/mtc.2003.175. PMID 12771874
- [Background] Murtuza B, Pepper JR, Stanbridge RD, Darzi A, Athanasiou T. Does minimal-access aortic valve replacement reduce the incidence of postoperative atrial fibrillation? Tex Heart Inst J. 2008;35(4):428-38. PMID 19156237
- [Background] Kuhn-Regnier F, Natour E, Dhein S, Dapunt O, Geissler HJ, LaRose K, Gorg C, Mehlhorn U. Beta-blockade versus Buckberg blood-cardioplegia in coronary bypass operation. Eur J Cardiothorac Surg. 1999 Jan;15(1):67-74. doi: 10.1016/s1010-7940(98)00289-9. PMID 10077376